CLINICAL TRIAL: NCT04428060
Title: Assessment of the Efficacy of Personalized Physiology-guided Resuscitation in Patients With Cardiac Arrest: The PERSEUS Pilot Randomized Trial
Brief Title: PERSEUS-PS Randomized Controlled Trial
Acronym: PERSEUS-PS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial prematurely terminated as a result of the COVID-19 pandemic.
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Chalkias, MD, PhD, Assistant Professor of Anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTHDA-AC02
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest With Successful Resuscitation
Keywords: Resuscitation; Cardiac arrest; Physiology-guided treatment; Personalized treatment; Outcome; Physiology
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERSEUS CPR (Experimental): Patients will be resuscitated according to the PERSEUS protocol
  Interventions: Other: PERSEUS CPR
- CONTROL (Active Comparator): Patients will be resuscitated according to current Advanced Life Support guidelines
  Interventions: Other: Standard CPR

INTERVENTIONS:
Other: PERSEUS CPR — Resuscitation based on patient physiology
  Arms: PERSEUS CPR
Other: Standard CPR — Resuscitation based on current guidelines
  Arms: CONTROL

SUMMARY:
The PERSEUS protocol is a new approach to the resuscitation of highly monitored patients with cardiac arrest. It aims at the optimization of all the available physiological parameters and the full exploitation of both the "cardiac pump" and "thoracic pump'. This protocol will help to titrate chest compressions, ventilation, and vasopressor dosing to physiological parameters, increasing survival after cardiac arrest with favorable neurological outcome

DETAILED DESCRIPTION:
BACKGROUND

Since 2000, resuscitation guidelines remain uniform across all cardiac arrest patients, focusing on the delivery of chest compressions to a standardized rate and depth and algorithmic vasopressor dosing. Although the concept of goal-directed hemodynamic optimization as a treatment strategy to improve clinical outcome in critically ill patients has been tested since the 1980s, no human study has established that prospectively targeting hemodynamics during CPR improves outcomes until now. Nevertheless, individualizing resuscitation to the appropriate hemodynamic and ventilatory goals rather than a standard Bone-size-fits-all treatment seems a promising new therapeutic strategy that can be applied during resuscitation attempts in highly monitored patients.

The PERSEUS protocol is a new approach to the resuscitation of highly monitored patients with cardiac arrest. It has been developed based on our experience and the observation that the most important determinant of survival is the optimization of all the available physiological parameters and the full exploitation of both the "cardiac pump" and "thoracic pump'.

Physiological and pathophysiological aspects of cardiac arrest Cardiac arrest interval Immediately after the abrupt loss of effective blood flow, the hypotension-induced baroreflex withdrawal with the net increase in the vascular resistance maintains an impaired antegrade and pulmonary blood flow. The systemic and pulmonary blood flow continue for at least 30-60 s, until the pressure gradient between the aorta and the right side of the heart, as well as between the pulmonary artery and the left atrium, has been completely dissipated, resulting in a rapid increase in the volume of the right ventricle and the extrapericardial component of the pulmonary veins. When arterial and systemic venous pressures reach equilibrium, the mean systemic filling pressure (Pmsf) is approximately 6-12 mmHg. The coronary blood flow declines to zero, but CPP remains positive because of the retrograde coronary flow. However, this diminishes the removal of norepinephrine from the interstitial spaces, which together with the formation of cardiac edema prolongs vasoconstriction and enhances myocardial hypoperfusion and hypoxia.

At the same time, cerebral perfusion decreases while the damage of fatty acids of the neuronal cell membrane by reactive oxygen species leads to a progressive increase in membrane permeability and severe derangements of intracellular electrolytes, resulting in cell swelling and brain edema formation. This, together with venous congestion, increases intracranial pressure (ICP) and damages the neuropil and synaptic structures and/or contacts.

The PERSEUS personalized physiology-guided resuscitation protocol Recognizing cardiac arrest in highly monitored areas can be more difficult than in other hospital areas, such as the ward. Considering that the vast majority of alarms from sensors are false alarms, cardiac arrest should be recognized and confirmed by the combined assessment of the rhythm, the arterial blood pressure and waveform, the abrupt decrease of ETCO2, and the loss of carotid pulse. Once cardiac arrest is confirmed, CPR should be initiated without delay with high-quality chest compressions according to the recent resuscitation guidelines. However, the effectiveness of chest compressions is depending on the venous return, which is proportional to the pressure gradient between Pmsf and CVP, and particular attention is needed by the rescuers to determine Pmsf within the first 5-7.5 s of cardiac arrest and prior to the onset of chest compressions. The Pmsf is a quantitative measurement of the patient's volume status and represents the tone of venous reservoir, indicating the pre-arrest "vasoreactivity" status of the patients. Therefore, optimizing Pmsf during CPR is paramount for increasing survival rates.

During the first cycle of CPR, the resuscitation efforts must maintain a relaxation DAP of ≥ 40 mmHg (calculated at the time of full chest decompression). In patients with a lower DAP, administration of epinephrine or vasopressin should be based on the pre-arrest value of Pmsf and/or systemic vascular resistance (SVR) and is anticipated to be beneficial in those with Pmsf < 6 mmHg and/or SVR < 800 dynes·sec·cm-5, enhancing volume recruitment from the unstressed compartment and increasing the stressed volume. In all other patients, the vasoreactivity will be maintained for some time provided that intravascular volume and chest compressions are sufficient. Therefore, circulatory volume should be increased in patients with a pre-arrest CVP < 2 mmHg using a fluid bolus and/or the passive leg-raising maneuver. However, it should be noted that rapid and liberal fluid administration during CPR may lead to an excessive increase in RAP, aggravating venous return and CPP, especially when administered via a jugular or subclavian central venous catheter. At the onset of cardiac arrest, ventilatory parameters should be changed to tidal volume 6 ml/kg, respiratory rate 10 min-1, I:E 1:2, PEEP 0 cm H20, and FiO2 100%. During this cycle, all other treatment efforts must follow current recommendations for standard CPR.

After the onset of the second cycle of CPR, the resuscitation efforts should be continued as above while assessing ETCO2. As stated previously, ventilation during CPR by using currently recommended chest compression rates may take place entirely below functional residual capacity and may not provide adequate blood oxygenation due to small airway closure, increasing pulmonary vascular resistance and impairing gas exchange. Therefore, mean airway pressure should be maintained 40-45 cmH2O in patients with DAP ≥ 40 mmHg and ETCO2 < 10 mmHg to facilitate gas exchange. On the contrary, all patients with DAP > 40 mmHg and ETCO2 > 15 mmHg should be assessed for hypercapnia, and if present, they should be treated by increasing the ventilatory rate by up to 50% (or less if necessary to maintain DAP ≥ 40 mmHg). Also, severe acidosis should be treated immediately because it causes vasodilatation which may decrease venous return and CPP.

During the third cycle of CPR, the resuscitation efforts should be continued as above while assessing ScvO2, which should be maintained 65-80%. In patients with ScvO2 < 65%, transfusion of red blood cells should be initiated when Hb is ≤8 g/dl to improve oxygen delivery. In patients with Hb > 8 g/dl, a fluid bolus should be given to improve circulatory flow provided that DAP is maintained ≥ 40 mmHg. In patients with DAP ≥ 40 mmHg and a ScvO2 value of > 80%, hypothermia should be excluded and treated aggressively if present, the FiO2 should be decreased in case of hyperoxemia (PaO2 > 200 mmHg), and a low-dose vasodilator may be considered when microcirculatory shunting and loss of hemodynamic coherence between macro- and microcirculation can be directly assessed or possible (e.g., DAP ≥ 40 mmHg, Hb > 8 g/dl, PaO2 > 200 mmHg, ScvO2 > 80%, and mixed venous oxygen tension ≤ 26 mmHg (if available), with or without hyperlactatemia). In patients with normal ScvO2, trend cerebral oxygenation monitoring (near-infrared spectroscopy - NIRS) should be used because it focuses more on the amount of change from the pre-arrest baseline cerebral oxygenation value. Decreasing FiO2 until PaO2 is 200 mmHg can be considered when NIRS is > 50% of the prearrest value, while HUP-CPR (30°) should be considered in patients with NIRS ≤ 30% of the pre-arrest value and signs or known increased intracranial pressure. The resuscitation efforts may be considered as adequate in patients who have reached the pre-defined targets and have a NIRS of 30-50% of the pre-arrest value, and should be continued by repeating the approach from the beginning.

AIM

The PERSEUS resuscitation protocol is a new approach to the resuscitation of highly monitored patients with cardiac arrest and may help to titrate chest compressions, ventilation, and vasopressor dosing to physiological parameters. The aim of this double-center study is to investigate if resuscitation with the PERSEUS protocol can increase survival after cardiac arrest with favorable neurological outcome.

METHODS

Design This is a prospective observational study designed in accordance with the declaration of Helsinki. The study will be register at Clinical Trials.gov and has been approved by the Institutional Review Board of the University Hospital of Larisa, under the reference number 2670/3-2-2020.

Patient eligibility All intubated and mechanically ventilated adult patients (≥ 18 years of age) with a CPR event requiring chest compressions in a highly monitored area [Operating Room, Intensive Care Unit (ICU), or Emergency Department] will be eligible for inclusion. Each patient will be allocated into two groups; patients in group A will be resuscitated with the PERSEUS protocol, while patients in group B will receive standard CPR according to the latest European Resuscitation Council guidelines on resuscitation. Random allocation will be carried out by a researcher who will not be involved in data collection using the sealed envelope technique.

Data Collection and Monitoring Data analysis will be based on predefined data points on a prospective data collection form. The staff will be blinded to measurements until the end of the study and all data are analyzed. Clinical monitoring throughout the study will be performed to maximize protocol adherence, while an independent Data and Safety Monitoring research staff will monitor safety, ethical, and scientific aspects of the study.

We will use the Utstein-style templates for in-hospital cardiac arrest data. Return of spontaneous circulation will be defined for all rhythms as the restoration of a spontaneous perfusing rhythm for more than 20 minutes. Survival with a favorable neurological outcome will be defined as a cerebral performance category (CPC) score of 1, 2 or no change from baseline. The CPC scoring system assesses functional outcomes among survivors of cardiac arrest and has been extensively validated and shown to reliably predict functional neurological disability.

Data management The goal of the clinical data management plan is to provide high-quality data by adopting standardized procedures to minimize the number of errors and missing data, and consequently, to generate an accurate database for analysis. Remote monitoring is performed to signal early aberrant patterns, issues with consistency, credibility and other anomalies. Any missing and outlier data values will individually revised and completed or corrected whenever possible.

Ethics and dissemination The study will be performed according to national and international guidelines. The present research investigation was reviewed by the IRB at the Larisa University Hospital and determined to be IRB exempt.

Competing interests None declared.

ELIGIBILITY:
Inclusion Criteria:

* invasive arterial blood pressure monitoring prior to and during CPR
* first compression of CPR captured on transmitted arterial blood pressure waveform data
* internal jugular or subclavian central venous catheter prior to and during CPR
* patients with measurement of systemic vascular resistance prior to and during CPR

Exclusion Criteria:

* unable to determine any of the aforementioned parameters during CPR
* unable to determine when CPR started and stopped
* subjects within the exclusion period of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
ROSC | From start of CPR until return of spontaneous circulation, assessed up to 60 minutes
  Return of spontaneous circulation

SECONDARY OUTCOMES:
ICU length of stay | Up to 8 weeks
  Days hospitalized in the intensive care unit
Days on mechanical ventilation | Up to 8 weeks
  How many days the patient will be mechanically ventilated
Survival to hospital discharge | Up to 8 weeks
  Dead or alive at hospital discharge with favorable neurological outcome (CPC 1 or 2)
1-month survival | At 1 month after hopsital discharge
  Dead or alive at 1 month after hospital discharge with favorable neurological outcome (CPC 1 or 2)
3-month survival | At 3 months after hopsital discharge
  Dead or alive at 3 months after hospital discharge with favorable neurological outcome (CPC 1 or 2)

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Chalkias, MD, PhD, Principal Investigator — University of Thessaly
Locations (1):
- University Hospital of Larisa, Department of Anesthesiology, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No
PD may be shared with other researchers upon reasonable request

REFERENCES:
- [Background] Sutton RM, French B, Meaney PA, Topjian AA, Parshuram CS, Edelson DP, Schexnayder S, Abella BS, Merchant RM, Bembea M, Berg RA, Nadkarni VM; American Heart Association's Get With The Guidelines-Resuscitation Investigators. Physiologic monitoring of CPR quality during adult cardiac arrest: A propensity-matched cohort study. Resuscitation. 2016 Sep;106:76-82. doi: 10.1016/j.resuscitation.2016.06.018. Epub 2016 Jun 24. PMID 27350369
- [Background] Jellinek H, Krenn H, Oczenski W, Veit F, Schwarz S, Fitzgerald RD. Influence of positive airway pressure on the pressure gradient for venous return in humans. J Appl Physiol (1985). 2000 Mar;88(3):926-32. doi: 10.1152/jappl.2000.88.3.926. PMID 10710387
- [Background] Aya HD, Cecconi M. Can (and should) the venous tone be monitored at the bedside? Curr Opin Crit Care. 2015 Jun;21(3):240-4. doi: 10.1097/MCC.0000000000000199. PMID 25887298
- [Background] Berg RA, Sutton RM, Reeder RW, Berger JT, Newth CJ, Carcillo JA, McQuillen PS, Meert KL, Yates AR, Harrison RE, Moler FW, Pollack MM, Carpenter TC, Wessel DL, Jenkins TL, Notterman DA, Holubkov R, Tamburro RF, Dean JM, Nadkarni VM; Eunice Kennedy Shriver National Institute of Child Health and Human Development Collaborative Pediatric Critical Care Research Network (CPCCRN) PICqCPR (Pediatric Intensive Care Quality of Cardio-Pulmonary Resuscitation) Investigators. Association Between Diastolic Blood Pressure During Pediatric In-Hospital Cardiopulmonary Resuscitation and Survival. Circulation. 2018 Apr 24;137(17):1784-1795. doi: 10.1161/CIRCULATIONAHA.117.032270. Epub 2017 Dec 26. PMID 29279413
- [Background] Chalkias A, Xanthos T. Timing positive-pressure ventilation during chest compression: the key to improving the thoracic pump? Eur Heart J Acute Cardiovasc Care. 2015 Feb;4(1):24-7. doi: 10.1177/2048872613516923. Epub 2013 Dec 12. PMID 24381094
- [Background] Chalkias A, Pavlopoulos F, Koutsovasilis A, d'Aloja E, Xanthos T. Airway pressure and outcome of out-of-hospital cardiac arrest: A prospective observational study. Resuscitation. 2017 Jan;110:101-106. doi: 10.1016/j.resuscitation.2016.10.023. Epub 2016 Nov 10. PMID 27840003
- [Background] Chalkias A, Arnaoutoglou E, Xanthos T. Personalized physiology-guided resuscitation in highly monitored patients with cardiac arrest-the PERSEUS resuscitation protocol. Heart Fail Rev. 2019 Jul;24(4):473-480. doi: 10.1007/s10741-019-09772-7. PMID 30741366